CLINICAL TRIAL: NCT03721016
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of MT10109L (NivobotulinumtoxinA) for the Treatment of Glabellar Lines With or Without Concurrent Treatment of Lateral Canthal Lines
Brief Title: MT10109L in the Treatment of Glabellar Lines (GL) With or Without Concurrent Treatment of Lateral Canthal Lines (LCL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT10109L-005; 2014-005301-21 (EudraCT Number)
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Glabellar Lines; Lateral Canthal Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MT10109L Dose 1 + Placebo (Experimental): MT10109L Dose 1 will be injected into the Glabellar Lines (GL) and Placebo into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  Interventions: Drug: MT10109L; Drug: Placebo
- MT10109L Dose 1 + MT10109L Dose 2 (Experimental): MT10109L Dose 1 will be injected into the Glabellar Lines (GL) and MT10109L Dose 2 into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  Interventions: Drug: MT10109L
- Placebo (Placebo Comparator): Placebo will be injected into the Glabellar Lines (GL) and into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT10109L — MT10109Lwill be injected into either the Glabellar Lines (GL), Lateral Canthal Lines (LCL), or both.
  Other Names: NivobotulinumtoxinA
  Arms: MT10109L Dose 1 + MT10109L Dose 2; MT10109L Dose 1 + Placebo
Drug: Placebo — Placebo will be injected into either the Glabellar Lines (GL), Lateral Canthal Lines (LCL), or both.
  Arms: MT10109L Dose 1 + Placebo; Placebo

SUMMARY:
To evaluate the safety and efficacy of MT10109L for the treatment of glabellar lines (GL) with or without concurrent treatment of lateral canthal lines (LCL) in participants with moderate to severe GL and LCL.

ELIGIBILITY:
Inclusion Criteria

• Female participants must not be pregnant or planning to get pregnant and willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period.

Exclusion Criteria

* Known immunization or hypersensitivity to any botulinum toxin serotype.
* Any medical condition that may put the participant at increased risk with exposure to MT10109L including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* History of facial nerve palsy.
* Any uncontrolled systemic disease.
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study intervention).
* Anticipated need for surgery or overnight hospitalization during the study.
* Prior exposure to botulinum toxin of any serotype for any reason.
* Prior periorbital surgery, facial lift (full face or mid-face), thread lift, brow lift, or related procedures (eg, eyelid [blepharoplasty] and/or eyebrow surgery).
* Prior facial treatment with permanent soft tissue fillers, synthetic implantation (eg, Gore-Tex®), and/or autologous fat transplantation.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Females who are pregnant, nursing, or planning a pregnancy during the study.
* Participants who plan for an extended absence away from the immediate area of the study site that would preclude them from returning for all protocol-specified study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SangMi Park, Study Director — Medytox Inc
Locations (21):
- United States (9):
  - Advanced Research Associates, Glendale, Arizona
  - Eye Research Foundation, Newport Beach, California
  - Skin Research Institute LLC, Coral Gables, Florida
  - Coleman Center for Cosmetic Dermatologic Surgery, Metairie, Louisiana
  - MD Laser, Skin, & Vein Institute, Hunt Valley, Maryland
  - Laser & Skin Surgery Center of New York, New York, New York
  - Bellaire Dermatology Associates, Bellaire, Texas
  - SkinDC, Arlington, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (4):
  - Dr. Shannon Humphrey Inc., Vancouver, British Columbia
  - Project Skin MD, Vancouver, British Columbia
  - Sweat Clinics of Canada, Toronto, Ontario
  - Bertucci MedSpa Inc., Woodbridge, Ontario
- Germany (4):
  - Studienzentrum Theatiner46, Munich, Bavaria
  - DRK-Kliniken Nordhessen, Kassel, Hesse
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf, North Rhine-Westphalia
  - RZANY & HUND - Privatpraxis fur Dermatologie und Asthetische Medizin, Berlin
- United Kingdom (4):
  - Saleh Aesthetic Clinic Ltd., Cheadle, England
  - Cranley Clinic, London, England
  - Bermuda Practice, Basingstoke, Hampshire
  - Meyer Clinic, Chichester, West Sussex

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 415 met the inclusion/exclusion criteria and were randomized.
Groups:
- Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL): Placebo was injected into the GL and into the LCL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into and Lateral Canthal Lines (LCL): MT10109L Dose 1 was injected into the GL and Placebo into the LCL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL): MT10109L Dose 1 was injected into the GL and MT10109L Dose 2 into the LCL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
Period: Overall Study
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Started | 82 | 173 | 160
Completed | 66 | 141 | 133
Not Completed | 16 | 32 | 27
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 16 | 13
Not completed — Lost to Follow-up | 4 | 6 | 5
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Site terminated by sponsor | 3 | 7 | 6
Not completed — Subject exited early due to COVID-19 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 415 participants included in the Intent To Treat (ITT) population (160 participants in the MT10109L Dose 1+2 group, 173 participants in the MT10109L Dose 1 group, and 82 participants in the placebo group).
Groups:
- MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL): MT10109L Dose 1 was injected into the GL and Placebo into the LCL: initial double-blind treatment on Day 1, and up to 2 additional blinded treatments during the retreatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL) | Total
Number analyzed (Participants) | 82 | 173 | 160 | 415
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 78 | 160 | 156 | 394
  >=65 years | 4 | 13 | 4 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (10.91) | 47.5 (11.49) | 46.2 (11.15) | 47 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 148 | 143 | 363
  Male | 10 | 25 | 17 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 25 | 28 | 66
  Not Hispanic or Latino | 69 | 148 | 132 | 349
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 2 | 3 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 1 | 2 | 6
  White | 75 | 168 | 151 | 394
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the Facial Wrinkle Scale With Photonumeric Guide (FWS)
Description: The outcome measured is the percentage of participants with a ≥ 2-grade improvement from baseline on the Facial Wrinkle Scale With Photonumeric Guide (FWS) according to investigator and participant assessments of Glabellar Lines (GL) severity at maximum frown at Day 30.
  The investigator and participant evaluates the participant's GL severity using a Facial Wrinkle Scale With Photonumeric Guide (FWS) at maximum frown on Day 30. The scale ranges from (0 to 3) where 0=none and 3 = severe.
Time Frame: Day 30
Population: All primary and secondary efficacy analyses endpoints were carried out using the Intent To Treat (ITT) analysis set, which was defined as all participants who were randomized. Multiple imputation method was used for missing variables in primary efficacy endpoint. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 82 | 173 | 160
Participants | 0 | 78 | 66

2. Secondary Outcome: The Duration of Glabellar Line (GL) Treatment in Participants Who Achieved a Rating of ≥ 2-grade Improvement From Baseline in GL Severity at Maximum Frown at Day 30 According to Investigator Assessments Using the Facial Wrinkle Scale (FWS)
Description: The investigator evaluates the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe. The outcome is measured as median time to loss of treatment effect (ie, return to moderate or severe GL severity at maximum frown using the FWS).
Time Frame: Day 1 (first treatment) to Day 180
Population: The analysis population for this outcome includes the participants who achieved a rating of ≥ 2-grade improvement from baseline in GL severity at maximum frown at Day 30 according to investigator assessments using the Facial Wrinkle Scale (FWS). This corresponds to the responders for Outcome 3. NA means no participant from the group achieved a rating of ≥ 2-grade improvement from baseline in GL severity. Note: Analyses of the secondary efficacy variables were performed using observed data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 0 | 83 | 83
days |  | 116.0 [92 to 128] | 118.0 [94 to 132]

3. Secondary Outcome: The Percentage of Responders for Investigator Assessments of Glabellar Lines (GL) Severity at Maximum Frown Using the Facial Wrinkle Scale (FWS)
Description: The percentage of Responders for Investigator Assessments of Glabellar Lines (GL) Severity at Maximum Frown Using the Facial Wrinkle Scale (FWS), where a Responder was defined as Achieving a ≥2-grade Improvement from Baseline at Maximum Frown at Day 30.
  The investigator evaluates the participant's GL severity using a 4-point scale (0 to 3) where 0=none and 3=severe.
Time Frame: Day 30
Population: All secondary efficacy analyses were carried out using the Intent To Treat (ITT) analysis set, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 81 | 163 | 154
Participants | 0 | 83 | 83

4. Secondary Outcome: The Percentage of Participants Reporting Mostly Satisfied/Very Satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 for Glabellar Lines (GL)
Description: The Satisfaction Question 5 grades facial line treatment satisfaction on a 5-point scale (-2 to 2) where -2=Very dissatisfied and 2=Very satisfied.
Time Frame: Day 60
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 74 | 159 | 150
Participants | 4 | 116 | 118

5. Secondary Outcome: The Percentage of Responders for Investigator Assessments of Glabellar Lines (GL) Severity at Rest Using the Facial Wrinkle Scale (FWS)
Description: The outcome was measured Among Participants Who Were Rated At least Mild at Rest at Baseline, where a Responder was Defined as Achieving a ≥1-grade Improvement from Baseline at Day 30
  The investigator evaluates the participant's GL severity using a 4-point scale (0 to 3) where 0=none and 3=severe.
Time Frame: Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 76 | 152 | 140
Participants | 11 | 84 | 100

6. Secondary Outcome: Secondary Safety: Number of Patients Who Experienced an Adverse Event (AE)
Description: This section focuses primarily on Treatment Emergent Adverse Events (TEAEs), i.e., AEs that started or worsened after the first dose of study intervention (Day 1) until up to 30 days after their last visit or study exit. The safety analyses were conducted in the Safety population. Unless otherwise noted, safety results refer to TEAEs.
Time Frame: The time frame for AEs is after the first dose (Day 1) and up to 30 days after their last visit or study exit (Day 360 unless participant exits earlier)
Population: All safety analyses were carried out using the Safety population, defined as participants who received at least 1 dose of study intervention. Participants were grouped based on their actual treatment received and not planned treatment. NOTE - 1 Participant randomized to 'Dose1 + Dose2' actually received treatment in the 'Dose1 + Placebo'. Therefore, the total number of participants analyzed in the 'MT10109L Dose 1 into GL + Placebo into LCL' arm is 174 instead of 173 that started in this arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 82 | 174 | 159
Participants | 31 | 82 | 61

7. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (BP)
Description: Changes in vital signs: Systolic BP
Time Frame: Baseline to Day 360 (Study exit)
Population: All safety analyses were carried out using the Safety population, which was defined as all participants who received at least 1 dose of study intervention. In Safety population, participants were grouped based on their actual treatment received and not planned treatment. In order to calculate the mean change from baseline, participants with non-missing analysis values at both baseline and post-baseline (Day 360) during that analysis visit were used.
Measure: Mean (Standard Deviation); unit: Change in mmHg
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 69 | 151 | 135
Change in mmHg | 2.5 (12.81) | 0 (12.33) | -1.7 (12.26)

8. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (BP)
Description: Changes in vital signs: Diastolic BP
Time Frame: Baseline to Day 360 (Study exit)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change in mmHg
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 69 | 151 | 135
Change in mmHg | -1.4 (7.81) | -0.9 (10.07) | -0.8 (8.64)

9. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: Changes in vital signs: Pulse Rate
Time Frame: Baseline to Day 360 (Study exit)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change in beats/min
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 69 | 151 | 135
Change in beats/min | -1.7 (11.25) | -1 (10.3) | -1 (8.93)

10. Secondary Outcome: Mean Change From Baseline in Respiratory Rate
Description: Changes in vital signs: Respiratory Rate
Time Frame: Baseline to Day 360 (Study exit)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change in breaths/min
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 69 | 151 | 135
Change in breaths/min | 0 (2.13) | 0.1 (2.28) | -0.2 (2.21)

11. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - Heart Rate
Description: Change from baseline for ECG safety population - Heart Rate
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in beats/min
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 134
Change from baseline in beats/min | 3.6 (9.79) | 2.4 (8.41) | 3.4 (9.51)

12. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - PR Interval
Description: Change from baseline for ECG safety population - PR Interval
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in msec
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 133
Change from baseline in msec | -3.2 (14.41) | -0.5 (12.41) | -0.7 (11.13)

13. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QRS Duration
Description: Change from baseline for ECG safety population - QRS duration
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in msec
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 134
Change from baseline in msec | 0.9 (5.78) | 1.1 (6.08) | 0.8 (6.06)

14. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QT Interval
Description: Change from baseline for ECG safety population - QT interval
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in msec
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 134
Change from baseline in msec | -10.4 (23.88) | -5.6 (21.0) | -8.0 (22.69)

15. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcB Interval
Description: Change from baseline for ECG safety population - QTcB interval
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in msec
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 134
Change from baseline in msec | 0.1 (15.5) | 1.2 (18.92) | 1.7 (17.65)

16. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcF Interval
Description: Change from baseline for ECG safety population - QTcF interval
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in msec
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 134
Change from baseline in msec | -3.5 (14.19) | -1.2 (15.91) | -1.8 (14.47)

17. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - RR Interval
Description: Change from baseline for ECG safety population - RR interval
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Change from baseline in msec
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 67 | 152 | 134
Change from baseline in msec | -46.0 (113.98) | -31.0 (113.11) | -44.6 (122.53)

18. Secondary Outcome: Number of Participants With Binding and Neutralizing Antibodies
Description: Only samples that tested positive in the binding antibody confirmatory assay were evaluated for neutralizing antibodies. The participants with positive neutralizing antibodies are only shown.
Time Frame: Day 360
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
Number analyzed (Participants) | 82 | 174 | 159
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: This section describes Treatment-Emergent Adverse Events (TEAEs) that started or worsened after the first dose of study intervention and within 30 days after the last visit or study exit (Day 360 unless the participant exits earlier)
Description: All safety analyses were carried out using the Safety population, defined as participants who received at least 1 dose of study intervention. Participants were grouped based on their actual treatment received and not planned treatment. NOTE - 1 Participant randomized to 'Dose1 + Dose2' actually received treatment in the 'Dose1 + Placebo'. Therefore, the total number of participants analyzed in the 'MT10109L Dose 1 into GL + Placebo into LCL' arm is 174 instead of 173 that started in this arm.
Arm/Group | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL)
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/174 | 0/159
Serious Adverse Events (participants affected / at risk) | 2/82 | 3/174 | 5/159
Other Adverse Events (participants affected / at risk) | 7/82 | 22/174 | 13/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) (N=82) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) (N=174) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL) (N=159)
Appendicitis (Infections and infestations) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Endometriosis [F] (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Into Both Glabellar Lines (GL) and Lateral Canthal Lines (LCL) (N=82) | MT10109L Dose 1 Into Glabellar Lines (GL) + Placebo Into Lateral Canthal Lines (LCL) (N=174) | MT10109L Dose 1 Into Glabellar Lines (GL)+ MT10109L Dose 2 Into Lateral Canthal Lines (LCL) (N=159)
Headache (Nervous system disorders) | 4 (4) | 14 (14) | 6 (6)
Injection site pain (General disorders) | 4 (4) | 9 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
General research agreement between the sponsor and PI's that includes a confidentiality section that includes a statement that the sponsor is and shall remain the exclusive owner of 'Information'. ) 'Information' shall include, but shall not be limited to, protocols, trade secrets, know-how, formulations, inventions, techniques, equipment, data and results.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03721016/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03721016/SAP_003.pdf